CLINICAL TRIAL: NCT06283147
Title: Risk Assessment and Management Program (RAMP) on Knee Osteoarthritis in Primary Care- a One-year Pragmatic Randomized Controlled Trial
Brief Title: Risk Assessment and Management Program (RAMP) on Knee Osteoarthritis in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Regina Wing Shan Sit, Professor Regina Wing Shan Sit, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023.530
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
Keywords: Risk assessment and Management Programme; Chronic Care Model
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Risk Assessment

STUDY DESIGN:
Intervention Model Description: The study is a 52-week, two-arm, parallel, doubled-blinded randomized clinical trial, evaluating the clinical efficacy of RAMP-Knee OA (N=114) versus usual care (N=114) on self-reported knee pain and other secondary outcomes.
Who Masked: Outcomes Assessor
Masking Description: All data collection will be performed by trained research assistants blinded to the allocation status of the patients, and statistician will analyse data without referring to allocation information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RAMP Knee OA (Experimental): Patients allocated to the intervention group will continue their "usual care" at the GOPCs, plus enrolment into the RAMP-Knee OA program.
  Interventions: Behavioral: Risk assessment and Management Programme - Knee Osteoarthritis
- Usual Care group (No Intervention): Patients allocated to the usual care arm will continue receiving their "usual care" at the GOPCs without any additional intervention. "Usual care" typically refers to the established and commonly provided treatments, interventions, and practices that patients would receive in routine clinical practice for their particular condition or disease. For GOPCs in Hong Kong, the follow-up period for all chronic diseases is typically every 4 months. Each consultation at GOPC has an average duration of 3-5 minutes, during which physicians will address all chronic diseases, including knee OA. Physicians may provide brief healthcare advice, prescribe chronic medications and analgesics if necessary, and refer patients to physiotherapy if indicated. The management approach for knee OA and other chronic diseases will be solely at the discretion of the attending physicians.

INTERVENTIONS:
Behavioral: Risk assessment and Management Programme - Knee Osteoarthritis — (i) Arthritis education: Topics will cover the 21 key messages identified in International Consensus List of Essential Statements for Osteoarthritis "What Do People With Knee or Hip Osteoarthritis Need to Know"
  (ii) Structured land-based exercise: We have selected strengthening, flexibility training (stretching), and aerobic exercise as our key components because they are most applicable in primary care settings.
  (iii) Weight Management: Weight management will be offered for participants with a BMI ≥ 23 kg/m2.
  (iv) Counselling support for psychosocial health: counselling support will be provided for those with mild to moderate anxiety and depression, insomnia and loneliness identified in the risk assessment.
  (v) Dietary advice: Online dietary education for musculoskeletal health (with reference to local context) will be provided. The dietitian will also provide support regarding specific dietary advice on weight management.
  Arms: RAMP Knee OA

SUMMARY:
The goal of this clinical trial is to determine the clinical effectiveness of a Chronic Care Model (CCM) named Risk Assessment and Management Program on Knee OA (RAMP-Knee OA) in adults with knee Osteoarthritis (Knee OA) at 52 weeks.

Participants will be screened for eligibility to participate. After confirming eligibility, participants will complete the baseline assessment and be randomized into one of the following groups (n=114 for each group):

1. RAMP Knee-OA group
2. Usual care group

Outcomes will be measured at baseline, week 16, week 32, and week 52.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine the clinical effectiveness of a Chronic Care Model (CCM) named Risk Assessment and Management Program on Knee OA (RAMP-Knee OA) in adults with knee Osteoarthritis (Knee OA) at 52 weeks. RAMP-knee OA is designed based on the validated framework of CCM, which identifies six important components including self-management support, clinical information systems, delivery system redesign, decision support, health care organization, and community resources.

The main questions the study aims to answer are:

In comparison with people undergoing usual care, whether:

* Participants in the RAMP-Knee OA group will report greater improvement in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain subscale
* Participants in the RAMP-Knee OA group will report greater improvement in physical function, self-management efficacy, lower limb muscle mass, psychosocial health, and quality of life

Participants will be screened for eligibility to participate. After confirming eligibility, participants will complete the baseline assessment and be randomized into one of the following groups (n=114 for each group):

1. RAMP Knee-OA group: Participants will be referred to the RAMP-Knee OA clinic operated by a Registered Nurse, which will be a face-to-face consultation scheduled every 4 months following patients' usual clinic appointments. A total of 4 sessions will be provided for each enrolled participant over one year. The content of the Programme centers around arthritis education, structure-land base exercise, and weight management, with the additional component of counseling support and dietary advice on musculoskeletal health.
2. Usual care group: Participants allocated to the usual care group will continue with their standard usual care (follow-up appointment at General Out Patient Clinic (GOPC) is typically every 4 months). The management approach for knee OA and other chronic diseases will be solely at the discretion of the attending physicians.

Outcomes will be measured at baseline, week 16, week 32, and week 52. Demographic data and knee pain duration will be collected at baseline assessment. Outcomes to measure include the severity of knee pain, physical function, level of physical activity, self-efficacy, level of anxiety and depression, insomnia, loneliness, health-related quality of life, and lower limb muscle mass. The use of co-intervention, analgesics, and other over-the-counter drugs will be recorded.

The baseline characteristics of the two groups will be compared using the independent samples t-test or the Mann-Whitney test for continuous variables and chi-square test for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Knee OA based on clinical criteria of the American Rheumatology College
* Moderate to severe Knee pain for 3 months or longer (average score of 4 or greater on a 0-10 pain scale in the past 3 months)

Exclusion Criteria:

* Participants with potential serious knee pathology (e.g. inflammatory arthritis, acute trauma, malignancy)
* Previous Knee replacement
* Scheduled knee joint replacement surgery within 1 year
* Participants who are unable to reliably participate (e.g. those who do not speak Chinese or unable to attend study intervention)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Knee pain | Baseline, week 16, week 32, week 52
  Knee pain as measured by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

SECONDARY OUTCOMES:
Physical Function | Baseline, week 16, week 32, week 52
  Physical function measured by WOMAC function subscale
Physical function | Baseline, week 16, week 32, week 52
  Physical function measured by 30-second chair and stand performance test
Lower limb muscle mass | Baseline, week 16, week 32, week 52
  Lower limb muscle mass measured by bio-impedance analysis
Level of physical activity | Baseline, week 16, week 32, week 52
  Level of physical activity measured by Chinese International Physical Activity Questionnaire (Short form)
Self-Management efficacy | Baseline, week 16, week 32, week 52
  Self-management efficacy measure by Pain-Self Efficacy questionnaire
Level of Anxiety | Baseline, week 16, week 32, week 52
  Anxiety measured by Generalized Anxiety Disorder -7
Level of Depression | Baseline, week 16, week 32, week 52
  Depression measured by Patient Health Questionnaire -9
Insomnia | Baseline, week 16, week 32, week 52
  Insomnia measured by 7 item Insomnia Severity Index
Loneliness | Baseline, week 16, week 32, week 52
  Loneliness measured by 6 item De Jong Gierveld Loneliness Scale
Health related Quality of Life | Baseline, week 16, week 32, week 52
  Health related Quality of life measured by Euroquol- 5D-5L
Demographic data | Baseline
  Demographic data such as height, weight, BMI, age, sex, knee pain duration, chronic comorbid conditions, chronic medications

CONTACTS AND LOCATIONS:
Overall Officials: Regina Wing Shan SIT, M.D., Principal Investigator — Jockey Club School of Public Health and Primary Care, Chinese University of Hong Kong
Locations (1):
- Lek Yuen GOPC, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sit RW, Yip BH, Choi SY, Wong MC, Law SW, Lam CY, Hunter D, Wong SY. Risk Assessment and Management Program (RAMP) on knee osteoarthritis in primary care-a one-year pragmatic randomized controlled trial. Trials. 2026 Feb 3. doi: 10.1186/s13063-026-09469-x. Online ahead of print. PMID 41629997